CLINICAL TRIAL: NCT00683293
Title: Laparoscopic Hysterectomy: a Clinical Randomized Trial Comparing Conventional and Robot-assisted(Da Vinci®)Techniques
Brief Title: Clinical Trial Comparing Conventional and Robot-assisted(Da Vinci®)Laparoscopic Interventions for Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dimitri Sarlos, Head Gynaecology and oncological Gynaecology, Kantonsspital Aarau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSA-RobHyst
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Laparoscopic Technique no Switch to Open; Duration of Surgery; Intraoperative Complications; Postoperative Complications
Keywords: Laparoscopic Hysterectomy; Robot-assisted Laparoscopic Hysterectomy; Robot-assisted Surgery
MeSH Terms: conditions — Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Randomized group of patients receiving conventional laparoscopic hysterectomy
  Interventions: Procedure: Conventional Laparoscopic Hysterectomy
- 2 (Active Comparator): Randomized group of patients receiving robot-assisted laparoscopic hysterectomy
  Interventions: Procedure: Robot-assisted (Da Vinci®) laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Conventional Laparoscopic Hysterectomy — Removal of uterus via standard laparoscopic techniques
  Other Names: - Minimal invasive hysterectomy,; - Laparoscopic removal of uterus,; - Minimal invasive removal of uterus
  Arms: 1
Procedure: Robot-assisted (Da Vinci®) laparoscopic hysterectomy — Removal of uterus by robot-assisted laparoscopic technique
  Other Names: - Robot-assisted(Da Vinci®)laparoscopic hysterectomy; - Robot-assisted minimal invasive hysterectomy
  Arms: 2

SUMMARY:
The aim of this study is to compare conventional with robot-assisted (Da Vinci®) laparoscopic hysterectomy regarding operating time peri-operative outcome and costs.

DETAILED DESCRIPTION:
During the last few years robot-assisted surgery has been introduced in many surgical specialties and experiences in gynaecological surgery are very limited.

Several aspects like the wider range of motion of robot-instruments leading to more precision in surgery, the 3 dimensional optical system and the ergonomically designed console may offer some advantages. For better judgment these possible benefits as well as safety and outcome need to be evaluated and compared with conventional laparoscopic hysterectomy techniques. This randomized clinical trail intends to compare conventional with robot-assisted(da Vinci®-System) laparoscopic hysterectomy regarding specific parameters. The focus of the study will be to investigate if the robot assisted procedure shows significant advantages for the patient considering duration of surgery, complications, hospitalisation and costs.

ELIGIBILITY:
Inclusion Criteria:

* Indication for laparoscopic hysterectomy
* Patients BMI < 40
* Signed consent

Exclusion Criteria:

* Estimated uterus weight >400 g
* No combination with other procedures
* No underlying malignant condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Sarlos, MD, Study Chair — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Switzerland

REFERENCES:
- [Result] Sarlos D, Kots L, Stevanovic N, von Felten S, Schar G. Robotic compared with conventional laparoscopic hysterectomy: a randomized controlled trial. Obstet Gynecol. 2012 Sep;120(3):604-11. doi: 10.1097/AOG.0b013e318265b61a. PMID 22914470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2008 to 2011 All patients were recruited from our clinic
Groups:
- 1 Conventional Laparoscopic Hysterectomy: Randomized group of patients receiving conventional laparoscopic hysterectomy
  Conventional Laparoscopic Hysterectomy : Removal of uterus via standard laparoscopic techniques
- 2 Robot-assisted Laparoscopic Hysterectomy: group of patients that receied robot-assisted laparoscopic hysterectomy Robot-assisted (Da Vinci®) laparoscopic hysterectomy : Removal of uterus by robot-assisted laparoscopic technique after randomization
Period: Overall Study
Arm/Group | 1 Conventional Laparoscopic Hysterectomy | 2 Robot-assisted Laparoscopic Hysterectomy
Started | 50 | 50
Completed | 48 | 47
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Conventional Laparoscopic Hysterectomy | 2 Robot-assisted Laparoscopic Hysterectomy | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (6) | 46.3 (4.2) | 46 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Duration of Surgery
Description: •Mean Time to complete surgery from cut to suture
Time Frame: after surgey
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1 Conventional Laparoscopic Hysterectomy | 2 Robot-assisted Laparoscopic Hysterectomy
Number analyzed (Participants) | 48 | 47
minutes | 75 (21) | 106 (29)

2. Secondary Outcome: Complications
Time Frame: up to 2 weeks
Measure: Number; unit: participants
Arm/Group | 1 Conventional Laparoscopic Hysterectomy | 2 Robot-assisted Laparoscopic Hysterectomy
Number analyzed (Participants) | 48 | 47
participants | 4 | 5

ADVERSE EVENTS:
Time Frame: 2008 to 2011
Arm/Group | 1 Conventional Laparoscopic Hysterectomy | 2 Robot-assisted Laparoscopic Hysterectomy
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes